CLINICAL TRIAL: NCT00085917
Title: A Randomized Controlled Trial to Evaluate the Safety and Efficacy of Twice-Weekly Peginterferon Alpha 2a and Ribavirin Induction Therapy for Chronic Hepatitis C in Patients Who Are Coinfected With HIV-1
Brief Title: Peginterferon Alpha-2a and Ribavirin to Treat Hepatitis C in HIV-infected Patients
Acronym: PIFNPK
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Shyamasundaran Kottilil, M.D./National Institute of Allergy and Infectious Diseases, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 040187; 04-I-0187
Record Dates: First submitted 2004-06-16; First posted 2004-06-17 (Estimated); Results first posted 2011-06-15 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Hepatitis C; HIV Infections
Keywords: Pegasys; Ribavirin; Early Virological Response; Hepatitis C; HIV
MeSH Terms: conditions — Hepatitis C; HIV Infections | interventions — peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard dose arm (Active Comparator): Pegylated interferon alfa -2a STANDARD DOSE Pegasys 180ug/week
  Interventions: Drug: standard dose pegylated interferon alfa -2a and ribavirin
- Double dose arm (Experimental): Double dose pegylated interferon with weight based Ribavirin
  Interventions: Drug: Double dose pegylated interferon with weight based Ribavirin

INTERVENTIONS:
Drug: Double dose pegylated interferon with weight based Ribavirin — pegylated interferon alfa -2a 180ug/twice weekly and weight based ribavirin for 4 weeks then pegylated interferon alfa -2a 180ug/ weekly for the remainder of the treatment
  Other Names: Pegasys
  Arms: Double dose arm
Drug: standard dose pegylated interferon alfa -2a and ribavirin — pegylated interferon alfa -2a 180ug weekly and weight based ribavirin for duration of the treatment
  Other Names: pegasys
  Arms: Standard dose arm

SUMMARY:
This study will evaluate the safety and effectiveness of combination therapy with peginterferon alpha-2a and ribavirin for treating hepatitis C virus (HCV) infection in HIV-infected patients. Peginterferon alpha with ribavirin is the therapy of choice for people with HCV alone. Peginterferon alpha-2a is a compound that results from attaching a polyethylene glycol molecule to interferon alpha-2a. This compound stays in the blood longer than unmodified interferon alpha-2a, causing a higher blood concentration and thus maintaining greater activity against the hepatitis C virus.

HIV-infected patients 18 years of age and older with chronic hepatitis C infection and a viral load greater than 2000 copies/mL may be eligible for this 2-1/2 year study. Candidates are screened with a medical history and physical examination, blood and urine tests, eye examination, chest x-ray, electrocardiogram (EKG), liver ultrasound, and pregnancy test in women who are able to become pregnant. If a recent liver biopsy is not available, this test is done to determine the type and severity of liver disease. The patient is given a sedative before the procedure. Then, the skin in the area over the biopsy site is numbed with a local anesthetic and a needle is inserted rapidly into and out of the liver to obtain a small tissue sample. The patient remains in the hospital overnight for monitoring.

Participants begin treatment with injections under the skin of peginterferon alpha-2a and ribavirin pills by mouth on study day 0. Peginterferon is given either once or twice a week for 4 weeks and then once a week for 44 weeks. Ribavirin is given daily. In addition, patients continue to take all other medications prescribed by their doctor. Clinic visits are scheduled for the following procedures:

* Days 1, 3, 4, 7, 10 and weeks 2, 3, and 4 - Blood tests for safety measures and to measure blood levels of HIV and HCV.
* Weeks 6, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 - Blood and urine tests to determine the side effects of treatment and its effect on the HCV infection. In addition, eye examinations are done every 3 months, and pregnancy and thyroid function tests are done several times during the treatment period.
* Week 48 or end of treatment - Treatment stops after 48 weeks. At this time, or earlier for those who do not complete the 48 weeks, patients return to the clinic for a chest x-ray, EKG, blood tests, and abdominal ultrasound. Patients are hospitalized for a repeat liver biopsy.
* Weeks 52, 56, 64 and 72 - Blood and urine tests to determine the side effects of treatment and its effect on the HCV infection, and a urine pregnancy test in women.

DETAILED DESCRIPTION:
Hepatitis C infection occurs in one-third of all HIV-infected individuals. Liver disease has become more significant among patients coinfected with HIV and HCV. Several studies have shown that coinfected individuals develop earlier and more severe liver disease. Pegylated interferon alpha with ribavirin has become the therapy of choice among people with HCV alone. This is a randomized controlled study to address the safety and efficacy of a 4 week induction therapy consisting of twice-weekly pegylated interferon alpha-2a and daily ribavirin on HIV-1 and hepatitis C coinfected individuals. Twenty-two patients who are infected with both HIV and HCV and who also have evidence of chronic hepatitis will be randomized to receive peginterferon alpha-2a either twice weekly or once weekly for four weeks. They will then continue with standard weekly peginterferon for 44 more weeks. The patients will receive standard daily dose of ribavirin during the entire 48 weeks. These patients will be monitored for peginterferon level, HCV viral load, HIV viral load and CD4 counts and undergo a baseline liver biopsy and another at the end of 72 weeks. The results of the study will enable us to better delineate the efficacy of twice weekly peginterferon induction therapy in suppressing the hepatitis C virus in the first 4 weeks of the therapy. Since viral suppression for hepatitis C in the early phase of the combination treatment has predictive values for long term eradication of the virus, a therapy that improves early viral suppression may improve the long term cure rate. This will be especially important given the current low cure rate of HCV among HIV coinfected individuals.

ELIGIBILITY:
INCLUSION CRITERIA

* Age greater than or equal to18 years.
* Documentation of HIV-1 infection by licensed ELISA test and confirmed by a Western Blot.
* Documentation of Hepatitis C infection by demonstration of a positive test for hepatitis C antibody and on HCV RNA level of 2000 or greater.
* Histopathologic features consistent with chronic hepatitis C on liver biopsy at the time of enrollment. A liver biopsy done for a subject within a year prior to his or her participation may be used as the baseline biopsy.
* Patients with CD4+ cell count greater than 200 cells/mm3 or CD4+ cell percentage greater than 14%.
* Ability to sign informed consent and willingness to comply with the study requirements and clinic policies.
* Serum phosphorus greater than or equal to 2.2 mg/dL and less than or equal to 4.4 (normal range NIH 2.3-4.3 mg/dL).
* Neutrophil count greater than or equal to 1000 cells/mm3.
* Platelets greater than or equal to 50,000/ mm3.
* Hemoglobin greater than or equal to 10.5 mg/dL.
* ALT less than 7 X the NIH upper limit of normal.
* Serum lipase less than 1.5 X the NIH upper limit of normal.
* Not pregnant or breast-feeding. Pregnancy test must be negative within two weeks prior to dosing with study medications.
* If the patient is able to become pregnant then she must use two effective methods of contraception during the study. Effective contraceptive methods include abstinence, surgical sterilization of either partner, barrier methods such as diaphragm, condom, cap or sponge, or use of hormonal contraception with an anti-HIV regimen that will not alter metabolism of hormonal contraception. This is advised on the basis of using ribavirin, which may have a potential teratogenic effect in pregnant women.
* Need to have a primary doctor outside of OP8 or as part of the OP8 training clinic who will be taking care of the patients for their HIV infection and liver disease.
* Willing to designate a person for durable power of attorney on the NIH form for medical research and medical care purposes at the NIH Clinical Center.
* Able to learn to safely inject medication subcutaneously or be able to find another person or a clinic to inject for him/her.

EXCLUSION CRITERIA

* Patient should not be on other experimental therapies during their participation in this protocol.
* Patients should not have used interferon or peginterferon previously for the treatment of hepatitis C
* Liver histology which, in the opinion of Clinical center pathologist, is consistent with any other co-existent cause of chronic liver disease as defined as chronic hepatitis B with positive HBSag, autoimmune hepatitis with a positive ANA greater than 1 unit or positive anti mitochondrial antibody greater than 1 unit, cholestatic disease with persistent elevation of Alkaline phosphatase, primary biliary cirrhosis or sclerosing cholangitis, Wilson's disease, alpha-1-antitrypsin deficiency, steatohepatitis (alcohol or non alcoholic) with marked steatosis, many Mallory bodies, or extensive zone 3 periportal fibrosis.
* Hemochromatosis or secondary iron overload as defined by (1) an elevated serum ferritin or an iron saturation (serum iron/IBC X 100%) of greater than 50% and (2) presence of 3+ or more stainable Iron on liver biopsy according to the study pathologist or a history of previous phlebotomy for Iron overload will undergo HFE genetic counseling and those with a positive HFE genetic test demonstrating homozygosity for C282Y and H63D are not eligible. Those who have compound heterozygosity to C282Y and H63D are also not eligible.
* Child Turcotte Pugh score greater than 7.
* PT-INR greater than 2 or history of hemophilia.
* Organ transplant recipient.
* Creatinine clearance less than 50 mL/min.
* Elevated alpha-fetoprotein level (greater than 100 ng/mL).
* Coexisting neoplastic disease except for Kaposi's Sarcoma, any non-metastatic skin cancer that has been resected, non-metastatic cervical or anal cancer that has been resected.
* Severe cardiac or pulmonary decompensation.
* Severe psychiatric disorder that would interfere with the adherence to protocol requirements.
* Preexisting autoimmune disorders including inflammatory bowel diseases, psoriasis, and optic neuritis.
* Preexisting uncontrolled seizure disorder.
* Preexisting pancreatitis.
* Severe retinopathy as determined by the ophthalmologist.
* Hemoglobinopathy.
* Currently taking didanosine as part of antiretroviral regimen.
* Direct bilirubin greater than 0.6 mg/dL.
* Using long-term systemic corticosteroids, immunosuppressives, or cytotoxic agents within 60 days of enrollment into the trial.
* Chronic viral hepatitis of any other etiology other than hepatitis C.
* Active systemic infections other than hepatitis C and HIV.
* Liver disease caused by reasons other than hepatitis C like HBV, HDV, Wilson's, hemochromatosis, autoimmune hepatitis (ANA greater than 1 unit) except history of drug-associated hepatitis with discontinuation of the causative agent.
* Hepatic mass suggestive of hepatocellular carcinoma as detected by ultrasound scan.
* Alcohol or substance abuse that potentially could interfere with patient compliance.
* History of esophageal varices.
* Any systemic illness that will make it unlikely that the subject will be able to return to NIH for the required study visits.
* Evidence of gastrointestinal malabsorption or chronic nausea or vomiting.
* Male partners of pregnant women.
* Pregnant women.
* Breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2004-06; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shyam Kottilil, Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Alter MJ, Mast EE. The epidemiology of viral hepatitis in the United States. Gastroenterol Clin North Am. 1994 Sep;23(3):437-55. PMID 7989088
- [Background] Seeff LB, Buskell-Bales Z, Wright EC, Durako SJ, Alter HJ, Iber FL, Hollinger FB, Gitnick G, Knodell RG, Perrillo RP, et al. Long-term mortality after transfusion-associated non-A, non-B hepatitis. The National Heart, Lung, and Blood Institute Study Group. N Engl J Med. 1992 Dec 31;327(27):1906-11. doi: 10.1056/NEJM199212313272703. PMID 1454085
- [Background] Koretz RL, Abbey H, Coleman E, Gitnick G. Non-A, non-B post-transfusion hepatitis. Looking back in the second decade. Ann Intern Med. 1993 Jul 15;119(2):110-5. doi: 10.7326/0003-4819-119-2-199307150-00003. PMID 8512159

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period was over a period of 3 yrs from 2004 - 2007. Participants were recruited and screened through the OP8 clinic of the NIAID.
Pre-assignment Details: There were no significant events or approaches following participant enrollment prior to group assignments.
  However if enrolled participants subsequently developed exclusion criteria such as active alcohol or drug abuse, they were excluded from the study.
Groups:
- Pegasys Single Dose: pegylated interferon alfa -2a 180 mcg/week and weight based Ribavirin (1000daily for weight<75kg, 1200mg daily for weight >75kg)
  - Treatment for 48 weeks
- Pegasys Double Dose: pegylated interferon alfa -2a 180 mcg/twice week and weight based Ribavirin (1000daily for weight<75kg, 1200mg daily for weight >75kg) for 4 weeks then pegylated interferon alfa -2a 180 mcg/week and weight based Ribavirin (1000daily for weight<75kg, 1200mg daily for weight >75kg) for 44 weeks
  - Total Treatment for 48 weeks
Period: Overall Study
Arm/Group | Pegasys Single Dose | Pegasys Double Dose
Started | 15 | 14
Completed | 11 | 11
Not Completed | 4 | 3
Not completed — Adverse Event | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pegasys Single Dose | Pegasys Double Dose | Total
Number analyzed (Participants) | 15 | 14 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 14 | 29
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 48 (6.402) | 46 (5.93) | 47 (6.109)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 11 | 10 | 21
Region of Enrollment [Number; unit: participants]
  United States | 15 | 14 | 29

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Sustained Virologic Response (SVR)
Description: SVR [ Sustained virological response] SVR was defined as HCV RNA levels below the limit of detection 24 weeks after the end of treatment.
Time Frame: 72 weeks
Measure: Number; unit: participants
Arm/Group | Pegasys Single Dose | Pegasys Double Dose
Number analyzed (Participants) | 11 | 11
participants | 11 | 11

2. Secondary Outcome: Number of Participants With Normalization of Liver Enzymes
Description: normalization of liver enzymes :Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) Alanine aminotransferase (ALT): Normal 6 - 41 U/L Aspartate aminotransferase (AST) : Normal 9 - 34 U/L
Time Frame: week 24, week 48, week 72
Measure: Number; unit: participants
Arm/Group | Pegasys Single Dose | Pegasys Double Dose
Number analyzed (Participants) | 11 | 11
participants | 11 | 11

3. Secondary Outcome: Number of Participants With Adverse Events
Description: Adverse Events
  - Anemia, Neutropenia and Psychiatric adverse events
Time Frame: 48 weeks
Measure: Number; unit: participants
Arm/Group | Pegasys Single Dose | Pegasys Double Dose
Number analyzed (Participants) | 11 | 11
participants | 11 | 11

ADVERSE EVENTS:
Time Frame: 2 YEARS
Arm/Group | Pegasys Single Dose | Pegasys Double Dose
Serious Adverse Events (participants affected / at risk) | 4/11 | 7/11
Other Adverse Events (participants affected / at risk) | 9/11 | 9/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pegasys Single Dose (N=11) | Pegasys Double Dose (N=11)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 6 (6)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pegasys Single Dose (N=11) | Pegasys Double Dose (N=11)
Anemia (Blood and lymphatic system disorders) | 6 (6) | 7 (7)
Depression/anxiety (Psychiatric disorders) | 6 (6) | 6 (6)
Neutropenia (Blood and lymphatic system disorders) | 9 (9) | 8 (9)
Fatigue (General disorders) | 2 (2) | 3 (3)
Weight loss (General disorders) | 2 (2) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4) | 4 (4)
Elevated transaminases (Hepatobiliary disorders) | 8 (8) | 6 (6)

LIMITATIONS AND CAVEATS:
Small number of enrolled participants

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes